CLINICAL TRIAL: NCT03316729
Title: Evaluation of Safety and Thrombolytic Effect of Ascending Doses of DS-9231 (TS23) in Subjects With Intermediate-risk (Sub-massive) Acute Pulmonary Embolism (PE)
Brief Title: DS-9231 in Intermediate-risk (Sub-massive) Acute Pulmonary Embolism (PE)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Product development cancelled.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DS9231-A-U201; 2017-000552-25 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Embolism
Keywords: Sub-massive acute pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Ascending doses in sequential cohorts (1-3) will be evaluated against placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-9231 (Experimental): In conjunction with standard of care, participants will receive an intravenous infusion delivering DS-9231 at ascending dose levels in Cohort 1, 2, and 3
  Interventions: Drug: DS-9231
- Placebo (Placebo Comparator): In conjunction with standard of care, participants will receive an intravenous infusion delivering only saline solution as matching placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-9231 — DS-9231 in saline solution for intravenous infusion
  Other Names: Investigational product
  Arms: DS-9231
Drug: Placebo — Placebo is matching saline solution for intravenous infusion
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate safety and initial effectiveness of DS-9231 when taken together with current standard of care. Evaluation will be done with low, medium and then high doses of DS-9231 versus placebo, in participants with medium-risk acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Had protocol-defined pulmonary embolism (PE)
* Has stable systolic blood pressure (SBP) >90 mm Hg
* Has evidence of right ventricular (RV) dysfunction
* Has executed informed consent

Exclusion Criteria:

* Has history or plans for thrombotic therapy outside protocol allowance
* Has other contraindications for participation
* Has laboratory results outside protocol-specified limits
* Is pregnant, nursing, and/or not willing or able to use protocol-defined contraceptives
* Has history or condition, or participated in another investigational study that (per protocol or in the opinion of the investigator) might compromise:

  1. the safety or well-being of the participant or the participant's offspring
  2. the safety of study staff
  3. the analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in total thrombus volume | Baseline, 48-96 hours after study drug administration
Percentage of participants with various gradations of decrease in total thrombus volume | Baseline, 48-96 hours after study drug administration
Number of participants with major or clinically relevant nonmajor bleeding | within 7 days after study drug administration
Number of participants with adverse events | within 30 days after study drug administration

SECONDARY OUTCOMES:
Percent change from baseline in total thrombus volume | Baseline, 30 days after study drug administration
Percentage of participants with with various gradations of decrease in total thrombus volume | 30 days after study drug administration
Percent change from baseline in RV/ left ventricle (LV) diameter ratio | Baseline, 48-96 hours and 30 days after study drug administration
Number of participants with PE-related deaths | within 30 days after study drug administration
Number of participants who died from any cause | within 30 days after study drug administration
Percentage of participants with clinical deterioration requiring additional rescue therapy for PE | within 30 days after study drug administration
Number of participants with with recurrent, objectively documented venous thromboembolism (VTE) | within 30 days after study drug administration
Participant-reported quality of life on a proprietary scale | Baseline, Day 30 after study drug administration
Number of participants with major or clinically relevant nonmajor bleeding | within 30 days after study drug administration
Number of participants re-hospitalized for any reason | within 30 days after study drug administration
Number of participants with non-bleeding adverse events (AEs) | within 30 days after study drug administration
Number of participants with anti-drug antibodies (ADAs) | within 30 days after study drug administration
Plasma concentration of DS-9231 | Baseline to 30 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/